CLINICAL TRIAL: NCT02497365
Title: Besifloxacin Ophthalmic Suspension in Patients With Bacterial Keratitis: A Prospective, Randomized Clinical Study
Brief Title: Besifloxacin in Bacterial Keratitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jean Deschenes, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPHTHO101
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Bacterial Keratitis
Keywords: keratits; besifloxacin
MeSH Terms: interventions — besifloxacin; Tobramycin; Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Besifloxacin (Experimental): Patients presenting with bacterial keratitis. These patients will be treated with besifloxacin ophthalmic suspesnion 0.6%, initially 6x a day and tapered down as the patient's condition improves based on the clinical judgement of the treating physician.
  Interventions: Drug: Besifloxacin
- Group B: Fortified Antibiotics (Active Comparator): Patients presenting with bacterial keratitis. These patients will be treated initially with fortified cefazolin and vancomycin drops every 1 hour around the clock (24hours) for a minimum of 48 hours, and will subsequently have their dosages tapered gradually by the treating physician as is the standard of care for bacterial keratitis.
  Interventions: Drug: Tobramycin and Cefazolin

INTERVENTIONS:
Drug: Besifloxacin
  Arms: Group A: Besifloxacin
Drug: Tobramycin and Cefazolin — Fortified Tobramycin and Cefazolin eye drops
  Arms: Group B: Fortified Antibiotics

SUMMARY:
This is a study comparing a new treatment for bacterial keratitis (also known as corneal ulcers) with the current standard of care. It is a randomized trial, and the investigators plan to test whether besifloxacin (a new antibiotic) in comparison to the current standard of treatment, fortified antibiotic drops (cefazolin and tobramycin).

DETAILED DESCRIPTION:
Hypothesis: patients with bacterial keratitis treated with besifloxacin ophthalmic suspension will have non inferior clinical outcomes as compared to those treated with fortified antibiotic drops (tobramycin and cefazolin)

Bacterial keratitis is a serious ocular problem that can, if not appropriately treated, lead to corneal scarring, perforation, endophthalmitis, and ultimately blindness. Current accepted treatment by some practitioners at a major academic center (McGill University Department of Ophthalmology) for corneal ulcers involves aggressive therapy with fortified antibiotics1, typically tobramycin (for gram negative coverage) and either vancomycin or cefazolin (for gram positive and/or MRSA coverage).

However, there are a number of problems with this treatment method. Patients must obtain the fortified antibiotics from specific pharmacies who must compound the preparations, increasing cost to the patient and potentially risk of contamination. The regimen typically involves every hour, round the clock dosing for at least the 48 hours, causing significant distress to patients (many of whom are eldery) and their families, as well as compliance issues. Finally, fortified antibiotics are toxic, by retarding the epithelial healing rate, as well as having conjunctival and corneal toxic effects.

The investigators' overall goal is to determine whether besifloxacin (at less frequent dosing than that used with fortified antibiotics) can be used safely and effectively in the treatment of bacterial keratitis. Previous studies have examined its effect on bacterial conjunctivitis, but not to the investigators' knowledge bacterial keratitis. However, as some clinicians are already using besifloxacin in this purpose, the investigators wish to examine the safety and efficacy of this.

If the investigators' study shows that besifloxacin is safe and effective in the treatment of bacterial keratitis, a new treatment option for bacterial keratitis may emerge.

The investigators therefore plan to conduct a randomized, open label trial enrolling patients newly diagnosed and not previously treated with bacterial keratitis. The patients will be randomized to receive either besifloxacin 6 x daily initially, or fortified antibiotics (cefazolin and tobramycin) every hour. The investigators will follow the patients closely to try to evaluate whether besifloxacin is an effective treatment for bacterial keratitis.

This is a randomized, single-center, two-arm, open-label study comparing a novel therapy, besofloxacin ophthalmic suspension, to traditional therapy of fortified cefazolin and tobramycin drops, in the treatment of bacterial keratitis.

Patients presenting with bacterial keratitis to the McGill Ophthalmology Center at 5252 Maissoneuve in Montreal, will be offered the opportunity by the resident and staff physician on call, to enroll in the study, with full discussion of risks and benefits as detailed above. Referrals will come from outpatient clinics and emergency departments as detailed above. The population of patients is expected to be outpatients, with a wide range of age groups >18 years old (no pediatrics as the study center does not see any pediatric age patients).

If patients choose not to enroll in the study, they will proceed to receive standard treatment at the center.

If patients choose to enroll in the study, the resident or staff on call, will, in consultation with the study investigators (Dr Jean Deschenes), use a pre-determined random number generator to randomize the patients to A) Besifloxacin arm, or B) Fortified Antibiotics arm.

At the first visit, a complete anterior ophthalmological exam will be performed, along with a detailed ophthalmic and medical history. Corneal scrapings will be performed (blood agar, chocolate agar, Sabaroud agar, slide mount for gram stain).

The participant will then be prescribed either Besifloxacin or Fortified Antibiotics (Cefazolin and Tobramycin) depending on their randomization. The participants will need to take the prescription to an outside pharmacy for purchase at their own cost of the medications. Suggested pharmacies will be made for the Fortified Antibiotics arm (as is standard of care due to the limited number of pharmacies that prepare the compounded drops).

Participants will be re-evaluated multiple times following initial presentation.

In each arm the medication will be tapered according to the clinical discretion of the treating physicians. In the besifloxacin arm, only besifloxacin will be used. In the fortified antibiotics arm, the fortified drops will be tapered and may be switched to another standard of care medication (moxifloxacin drops) as the bacterial keratitis improves as per the typical treatment regimen. Importantly, in this arm, the treatment will be carried out as normal standard of care for bacterial keratitis.

In the besifloxacin arm, if, at the visit on day 8, previous corneal bacterial cultures remain positive, the patient will be crossed over into the fortified antibiotic arm. Otherwise, crossover may occur only if there is significant clinical deterioration by the treating physician that requires urgent intervention.

The expected duration of each subject participation is 4 months. Study enrollment is expected to last for about 4 months as well.

ELIGIBILITY:
Inclusion Criteria:

* • Provide signed and dated informed consent form

  * Willing to comply with all study procedures and be available for the duration of the study
  * Male or female, aged 18 or older
  * Clinically diagnosed bacterial keratitis, with any size ulcer > 1mm.

Exclusion Criteria:

* • Previously treated for current episode of bacterial keratitis with an antibiotic drop

  * Corneal Ulcers <1mm
  * Known allergic reaction to components of the study products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09; Primary Completion 2019-06 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Time to microbial sterilization of the infected cornea | 2-14 days
  We will take repeat cultures and determine when no more bacteria can be cultured

SECONDARY OUTCOMES:
Time until closure of epithelial defect | 2-14 days
Final pinhole corrected visual acuity | 4 months
Final corneal scar size | 4 months
Severe adverse events: corneal perforation, endophthalmitis | 4 months
Time until clinical resolution as determined by physician | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- McGill Academic Eye Center, Montreal, Quebec, Canada